CLINICAL TRIAL: NCT01326871
Title: A Phase Ib/II Trial of ALT-801 in Combination With Cisplatin and Gemcitabine in Muscle Invasive or Metastatic Urothelial Cancer
Brief Title: A Study of ALT-801 in Combination With Cisplatin and Gemcitabine in Muscle Invasive or Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-01-10
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Transitional Cell Carcinoma of Bladder; Urethra Cancer; Ureter Cancer; Malignant Tumor of Renal Pelvis
Keywords: cancer; immunotherapy; immunochemotherapy; combinational therapy; targeted; metastatic; muscle invasive; interleukin-2; cisplatin; gemcitabine; antitumor; TCR; T-cell receptor; p53; p53 gene; p53 tumor supressor protein; urothelial cancer; bladder cancer; renal pelvis cancer; ureters cancer; urethra cancer; HLA-A2 positive; HLA-A*0201/p53 aa264-272; HLA complex; Muscle Invasive or Metastatic
MeSH Terms: conditions — Urethral Neoplasms; Ureteral Neoplasms; Neoplasms; Neoplasm Metastasis; Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; ALT-801

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ALT-801 0.04 mg/kg with Cisplatin and Gemcitabine (Experimental)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Biological: ALT-801
- ALT-801 0.06 mg/kg with Cisplatin and Gemcitabine (Experimental)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Biological: ALT-801
- ALT-801 0.06 mg/kg with Gemcitabine (Experimental)
  Interventions: Drug: Gemcitabine; Biological: ALT-801

INTERVENTIONS:
Drug: Cisplatin — Intravenous infusion; 3 initial treatment courses and an additional 3 maintenance courses for responders (maintenance revised for Phase II): on day 1 of each course (if given)
  Arms: ALT-801 0.04 mg/kg with Cisplatin and Gemcitabine; ALT-801 0.06 mg/kg with Cisplatin and Gemcitabine
Drug: Gemcitabine — Intravenous infusion; 3 initial treatment courses and an additional 3 maintenance courses for responders (maintenance revised for Phase II); on day 1 and 8 of each course
Biological: ALT-801 — Intravenous infusion; 3 initial treatment courses and an additional 3 maintenance courses for responders (maintenance revised for Phase II): on day 3, 5, 8, and 12 of each course
  Other Names: c264scTCR-IL2

SUMMARY:
This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-801 in a biochemotherapy regimen either containing cisplatin and gemcitabine or containing gemcitabine alone in patients who have muscle invasive or metastatic urothelial cancer of bladder, renal pelvis, ureters and urethra. The purpose of this study is to evaluate the safety, determine the maximum tolerated dose (MTD) and the recommended dose (RD), and assess the anti-tumor response of ALT-801 in combination with cisplatin and gemcitabine or ALT-801 in combination with gemcitabine alone. The pharmacokinetic profile of ALT-801 in combination with cisplatin and gemcitabine will also be assessed. The study includes a dose escalation phase (Phase Ib) and a dose expansion phase (Phase II). Phase II has two treatment groups, Expansion Group 1 and Expansion Group 2. Expansion Group 2 is for platinum-refractory patients, consisting of two treatment arms based on the patient's renal function. Patients will enroll to Expansion Group 2 after stage 1 of the Group 1 expansion is complete.

DETAILED DESCRIPTION:
Bladder cancer is the fourth most common malignancy in men and the ninth most common in women in the US, with an estimated 68,810 new cases and 14,070 deaths for the year 2008. Approximately 90% to 95% of newly diagnosed patients are with transitional cell carcinomas (TCC). Approximately 20% to 25% contain advanced (muscle invasive or metastatic) disease. Muscle invasive bladder cancer is life threatening. Clinical trials have demonstrated that TCC is a chemotherapy-sensitive malignancy. Most current cancer treatment strategies involve the use of chemotherapeutic or biological drugs that have a low therapeutic ratio. The limitations are a consequence of effects of the therapeutic drug on normal tissues. One approach to control systemic exposure effects is to target the drug itself into the site of the tumor. For example, antibodies have been developed for use as tumor targeting agents and have had success in the clinic. However, despite the promise of antibody-based immunotherapy, there are limitations with these class of reagents. Even so, immunotherapy remains a promising approach to treat cancer.

One strategy that has received attention is treatment with cytokines such as IL-2 to enhance anti-tumor immunity. IL-2 has stimulatory effects on a number of immune cell types including T and B cells, monocytes, macrophages, lymphokine-activated killer cells (LAK) and natural killer (NK) cells. Based on the ability of IL-2 to provide durable curative anti-tumor responses, systemic administration of IL-2 has been approved to treat patients with metastatic melanoma or renal carcinoma. Unfortunately, the considerable toxicity associated with this treatment makes it difficult to achieve an effective dose at the site of the tumor and limits the population that can be treated. Thus, there is critical need for innovative strategies that enhance the effects of IL-2, to reduce its toxicity without compromising the clinical benefit, and to treat other diagnoses.

The study drug, ALT-801, is a biologic compound of interleukin-2 (IL-2) genetically fused to a humanized soluble T-cell receptor directed against the p53-derived peptides expressed on tumor cells. The p53 protein is one of the most important factors that protects from developing cancer and is also one of the most frequently mutated genes in many cancers, which include muscle-invasive bladder cancer. For any given cancer type, p53 dysfunction generally correlates with poor prognosis versus other the same site-of-origin. In some tumors, p53 mutation and over-expression also is associated with resistance to chemotherapy. This study is to further evaluate whether directing IL-2 activity using ALT-801 to the patient's tumor sites that over-express p53 results in clinical benefits

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARATERISTICS:

* Muscle invasive or metastatic urothelial cancer of bladder, ureters, renal pelvis, and urethra
* Histologically or cytologically confirmed with a clinical plan that would potentially include cisplatin* plus gemcitabine systemic therapy or with disease refractory to a first-line platinum-based therapy (as defined in the protocol).

  * Does not apply to patients screened for Phase II expansion
* Surgically incurable

PRIOR/CONCURRENT THERAPY:

* No concurrent radiotherapy, other chemotherapy, or other immunotherapy
* Must have recovered from side effects of prior treatments
* If prior Proleukin® treatment, must have had a clinical benefit
* No use of other investigational agents within 30 days of start or concurrently

PATIENT CHARACTERISTICS:

Age

* ≥ 18 years

Performance Status

* ECOG 0 or 1

Bone Marrow Reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1,500/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 10g/dL

Renal Function

* Glomerular Filtration Rate (GFR):

  * ≥ 50mL/min/1.73m^2 for cisplatin-containing regimen
  * ≥ 40mL/min/1.73m^2 for non-cisplatin-containing regimen

Hepatic Function

* Total bilirubin ≤ 1.5 X ULN
* AST, ALT, ALP ≤ 2.5 X ULN, or ≤ 5.0 X ULN (if liver metastases exists)
* PT INR ≤ 1.5 X ULN

Cardiovascular

* No congestive heart failure < 6 months
* No unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias
* No NYHA Class > II CHF
* Normal cardiac stress test required for subjects who are ≥ 50 years old, or have a history of EKG abnormalities, or have symptoms of cardiac ischemia or arrhythmia
* No uncontrolled hypertension

Pulmonary

* Not receiving chronic medication for asthma
* Normal clinical assessment of pulmonary function

Hematologic

* No evidence of bleeding diathesis or coagulopathy

Other

* Negative serum pregnancy test if female and of childbearing potential
* No women who are pregnant or nursing
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No known autoimmune disease other than corrected hypothyroidism
* No known prior organ allograft or allogeneic transplantation
* Not HIV positive
* No active systemic infection requiring parenteral antibiotic therapy
* No ongoing systemic steroid therapy required
* No history or evidence of CNS disease (Controlled brain metastases treated with radiation therapy or surgery where the disease has been clinically stable for a period of a least 3 months before screening is allowed)
* No psychiatric illness/social situation
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* Must provide informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - UF Health Center at Orlando Health, Orlando, Florida
  - Martin Health System, Stuart, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Robert Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Fairway, Kansas
  - Karmanos Cancer Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - St. Luke's Hospital and Health Network, Easton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1b and Phase 2 subjects were combined by ALT-801 dose level and whether they received cisplatin or did not.
Period: Overall Study
Arm/Group | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Gemcitabine
Started | 3 | 49 | 16
Completed | 3 | 21 | 1
Not Completed | 0 | 28 | 15
Not completed — Major surgery | 0 | 1 | 0
Not completed — SAE and death | 0 | 2 | 0
Not completed — Physician decision and decreased performance status | 0 | 1 | 0
Not completed — Disease progression | 0 | 11 | 5
Not completed — Did not qualify or consent for repeat treatment | 0 | 1 | 0
Not completed — Subject decision to continue survival follow-up only | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — DLT | 0 | 2 | 0
Not completed — SAE, disease progression and subject decision | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Other | 0 | 3 | 0
Not completed — SAE and disease progression | 0 | 0 | 1
Not completed — SAE and physician decision | 0 | 0 | 1
Not completed — Did not qualify/consent for repeat treatment, subject decision to continue survival follow-up only | 0 | 0 | 1
Not completed — Did not qualify or consent for repeat treatment and disease progression | 0 | 0 | 1
Not completed — Physician decision, AEs and subject compliance | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — SAE | 0 | 0 | 1
Not completed — Disease progression and death | 0 | 0 | 1
Not completed — Subject decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Gemcitabine | Total
Number analyzed (Participants) | 3 | 49 | 16 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (2.1) | 63 (7.9) | 65 (9.7) | 63 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 6 | 15
  Male | 2 | 41 | 10 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 47 | 15 | 65
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 3 | 46 | 13 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Subjects with Muscle Invasive or Metastatic Urothelial Cancer [Count of Participants; unit: Participants] | 3 | 49 | 16 | 68

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and/or the Recommended Dose (RD) for Dose Expansion of ALT-801 in Combination With Cisplatin and Gemcitabine or ALT-801 in Combination With Gemcitabine Alone
Time Frame: 8 weeks
Measure: Number; unit: mg/kg Recommended Dose
Groups:
- ALT-801: 0.04 mg/kg, 0.06 mg/kg: Recommended dose is ALT-801 0.06 mg/kg
Arm/Group | ALT-801: 0.04 mg/kg, 0.06 mg/kg
Number analyzed (Participants) | 9
mg/kg Recommended Dose | 0.06

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of AEs that occur or worsen after the first dose of study treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Gemcitabine
Number analyzed (Participants) | 3 | 49 | 16
Participants | 3 | 49 | 16

3. Primary Outcome: Objective Response Rate in Treated Patients
Description: Objective response rate (ORR) is defined as confirmed complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors [RECIST V1.0]: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR.
Time Frame: 12 weeks
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Gemcitabine
Number analyzed (Participants) | 3 | 49 | 16
percentage of participants | 100 [29 to 100] | 47 [33 to 62] | 6 [0 to 30]

ADVERSE EVENTS:
Arm/Group | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine | ALT-801 0.06 mg/kg With Gemcitabine
All-Cause Mortality (participants affected / at risk) | 2/3 | 42/49 | 16/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 20/49 | 8/16
Other Adverse Events (participants affected / at risk) | 3/3 | 49/49 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine (N=3) | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine (N=49) | ALT-801 0.06 mg/kg With Gemcitabine (N=16)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Death (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 3 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALT-801 0.04 mg/kg With Cisplatin and Gemcitabine (N=3) | ALT-801 0.06 mg/kg With Cisplatin and Gemcitabine (N=49) | ALT-801 0.06 mg/kg With Gemcitabine (N=16)
Fatigue (General disorders) | 2 | 36 | 5
Chills (General disorders) | 1 | 24 | 7
Pyrexia (General disorders) | 2 | 23 | 5
Oedema peripheral (General disorders) | 1 | 15 | 1
Pain (General disorders) | 1 | 7 | 1
Influenza like illness (General disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 39 | 8
Vomiting (Gastrointestinal disorders) | 3 | 29 | 6
Constipation (Gastrointestinal disorders) | 2 | 19 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 19 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 3 | 42 | 9
Neutrophil count decreased (Investigations) | 3 | 28 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 17 | 5
Blood creatinine increased (Investigations) | 0 | 19 | 4
Alanine aminotransferase increased (Investigations) | 1 | 15 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 11 | 5
Lymphocyte count decreased (Investigations) | 1 | 11 | 4
White blood cell count decreased (Investigations) | 2 | 11 | 3
Weight decreased (Investigations) | 0 | 6 | 1
Weight increased (Investigations) | 1 | 3 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 2
International normalised ration increased (Investigations) | 0 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 26 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 20 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 15 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 15 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 20 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 13 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 12 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 8 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 5 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 30 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 17 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 18 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 18 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 8 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 8 | 0
Dizziness (Nervous system disorders) | 0 | 6 | 1
Paraesthesia (Nervous system disorders) | 0 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 9 | 7
Embolism (Vascular disorders) | 0 | 6 | 2
Hypertension (Vascular disorders) | 0 | 3 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 5 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 3 | 0
Skin infection (Infections and infestations) | 1 | 2 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1
Root canal infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 6 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 3 | 3
Haematuria (Renal and urinary disorders) | 0 | 4 | 2
Proteinuria (Renal and urinary disorders) | 0 | 4 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 7 | 2
Anxiety (Psychiatric disorders) | 0 | 4 | 3
Confusional state (Psychiatric disorders) | 0 | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 4 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 3 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT01326871/Prot_SAP_000.pdf